CLINICAL TRIAL: NCT06627959
Title: StatSeal vs Figure-of-Eight Suture for Vascular Closure in AF Ablation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 348992
Record Dates: First submitted 2024-10-01; First posted 2024-10-04 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation (AF); Vascular Access
Keywords: atrial fibrillation; vascular closure; Statseal
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Statseal (Active Comparator): This group shall receive the StatSeal device for vascular closure
  Interventions: Device: Statseal
- Figure of eight suture (Active Comparator): This group shall receive the figure of eight suture (attached to a three-way stopcock) for vascular closure
  Interventions: Device: Figure of eight suture

INTERVENTIONS:
Device: Statseal — This is a vascular closure device which works independently of the clotting cascade to seal access sites
  Arms: Statseal
Device: Figure of eight suture — The figure of eight suture is commonly used for vascular access closure
  Arms: Figure of eight suture

SUMMARY:
This study, titled aims to compare two vascular closure techniques after catheter ablation for atrial fibrillation (AF). Catheter ablation is a common procedure used to treat AF, but after the procedure, It is important to close the access site in the blood vessel to prevent bleeding. This study will evaluate whether the StatSeal device, a haemostatic disc, can help patients recover more quickly compared to the traditional figure-of-eight suture technique.

The primary objective of the study is to determine whether StatSeal reduces the time it takes for patients to start walking after the procedure (known as Time to Ambulation). Secondary objectives include comparing the time to complete haemostasis, discharge eligibility, incidence of adverse events, and patient comfort between the two techniques.

Participants in the study will be randomly assigned to receive either the StatSeal device or the figure-of-eight suture after their AF ablation procedure. The study will recruit 160 participants across multiple hospital sites, with 80 participants in each group. Both techniques are standard methods, and participants will be closely monitored for safety throughout the study.

By comparing these two closure techniques, the study aims to improve the recovery process for patients undergoing AF ablation and provide evidence on which method leads to better outcomes and patient experiences.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age >18
* Elective catheter ablation for atrial fibrillation using a 6 to 14 Fr inner diameter introducer sheath with a minimum of 1 and maximum of 3 femoral venous access sites
* Willing and able to give informed consent

Exclusion Criteria:

* Active systemic or cutaneous infection, or inflammation in vicinity of the groin
* Platelet count < 100,000 cells/mm3
* BMI > 45 kg/m2 or < 20 kg/m2
* Attempted femoral arterial access or inadvertent arterial puncture
* Procedural complications that interfered with routine recovery, ambulation, or discharge times
* Incorrect sheath placement
* Intraprocedural bleeding or thrombotic complications
* Access site-specific eligibility criteria to exclude problems with gaining access or location of sheath
* History of bleeding diathesis, coagulopathy, hypercoagulability, or thromboembolic events

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2025-01-03 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Time to ambulation (TTA) after sheath removal | 1 day
  Time to ambulation is defined as the elapsed time between removal of the final sheath and the moment when the patient can stand and walk 20 feet without evidence of venous re-bleeding from the femoral access site.

SECONDARY OUTCOMES:
Time to haemostasis | 1 day
  time elapsed between removal of the vascular sheath and first observed and confirmed venous haemostasis, for each access site
Time to discharge eligibility | 1 day
  time elapsed between removal of the final sheath and when the patient is eligible for hospital discharge based solely on the assessment of the access site, as determined by the medical team
Time to discharge | 1 day
  time elapsed between removal of the final sheath and when the patient was discharged from the institution
Incidence of major periprocedural adverse events | 1 day
  defined as adverse events until hospital discharge requiring medical intervention.
Incidence of major adverse events | 30 days
  Major adverse events are defined as complications requiring medical intervention or hospitalisation
Incidence of minor adverse events | 30 days
  Minor adverse events are defined as AEs not requiring medical intervention.
Comparison of EuroQol EQ-5D-5L | 30 days
  Comparison of EuroQol 5-level EQ-5D score. The score is made up of two parts: the EQ-5D descriptive system and the EQ visual analogue scale (EQ-VAS). The first part covers five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension offers five response options (no problems, slight problems, moderate problems, severe problems, and extreme problems), from which an EQ-5D index score is calculated, ranging from 0 (death) to 1 (perfect health). The EQ-VAS assesses an individual's self-perceived health for the day on a vertical scale from 0 (worst imaginable health) to 100 (best imaginable health), where participants mark their current health status.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - The Essex Cardiothoracic Centre, Basildon, Essex
  - East Sussex Healthcare NHS Trust, Eastbourne
  - Norfolk and Norwich University Hospital, Norwich

IPD SHARING:
Plan to Share IPD: No